CLINICAL TRIAL: NCT04114175
Title: The Effects of Spinal Stabilization Exercises on Energy Expenditure in Individuals With Transtibial Amputatıon
Brief Title: Spinal Stabilization Exercises in Individuals With Transtibial Amputatıon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Principal Investigator, Senay Cerezci Duygu, Research Assistant, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KA19/143
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Amputees; Exercise Training; Physiotherapy; Energy Metabolism
Keywords: amputees; rehabilitation; energy expenditure; deep muscles of the back

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): People with unilateral transtibial amputation. Participants will be provided from the sample group according to the randomization.
  Interventions: Other: Exercise BE
- Spinal Stabilization Group (Experimental): People with unilateral transtibial amputation. Participants will be provided from the sample group according to the randomization.
  Interventions: Other: Exercise BE+SS

INTERVENTIONS:
Other: Exercise BE — Basic exercises related to amputation will be applied
  Arms: Control Group
Other: Exercise BE+SS — Basic exercises related to amputation + Spinal stabilization exercises will be applied
  Arms: Spinal Stabilization Group

SUMMARY:
Lower extremity amputation causes rapid changes in musculoskeletal system. With the effect of these changes, the energy requirement for prosthetic ambulance is much higher than normal ambulance. Although methods such as the reduction of the segmental load of the prosthesis and the preference of the different prosthetic components for energy expenditure have been emphasized, the effect of exercise types has not been investigated in our knowledge. Therefore, the aim of the current study is to investigate the effect of spinal (Core) stabilization exercises on energy expenditure in combination with the classical physiotherapy program in patients with unilateral transtibial amputation. Individuals with transtibial amputation included in the study will be randomly divided into two groups. In group 1, basic exercises related to amputation will be applied for 8 weeks and in group 2 basic exercises with spinal stabilization exercises will be applied to the individuals. At the beginning and at the end of the exercise intervention, energy expenditure and exercise capacity will be evaluated by a portable exercise test device during '6 Minutes Step Test'; fatigue assessment will be done before and after 6 Minutes Step Test with 'Modified Borg Scale'; the strength of deep spinal muscles will be evaluated with 'Stabilizer'; dynamic balance and functional mobility will be evaluated by 'Timed Up & Go' Test; and the effect of the prosthesis on mobility will be evaluated by the sub-scale 'Mobility' of 'Prosthetic Evaluation Questionnaire'.

ELIGIBILITY:
Inclusion Criteria:

* Having unilateral transtibial amputation of at least 6 months in which the stump volume becomes stable,
* Being prosthetic users (For homogenization of the groups in terms of external support used, individuals with transitibial amputation included in the study should use total contact socket and carbon foot prosthesis systems - Pin System, Passive Vacuum System or Active Vacuum System),
* Having at least "four" quadriceps and hamstring muscle strength in the amputated limb according to Lovett's manual muscle test method.

Exclusion Criteria:

* Having any disadvantage about prosthetic device usage in terms of stump length, shape and edema,
* Having movement limitation,
* Having phantom pain in the stump,
* Having any discomfort or health problem (cardiopulmonary, neurological or orthopedic problems) that may affect gait other than amputation,
* Having multiple extremity loss.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Energy expenditure and exercise capacity | 6 minutes
  Assessement will be with the exercise tester (COSMED, Fitmate Pro, Rome, Italy) during the 6 Minute Step Test .

SECONDARY OUTCOMES:
Fatigue | 20 seconds
  Assessement will be with "Modified Borg Scale" after 6 Minute Step Test. Pariticipants were shown the Modified Borg Scale, which is a vertical scale from 0 to 10 in which numbers are anchored with corresponding verbal expressions of progressively increasing intensity. The patients were asked to rate their fatigue by selecting the number with the corresponding words that most appropriately described their sensation of fatigue. The minimum value that can be obtained as a result of the evaluation is 0 (Nothing at all), the maximum value is 10 (Maximal).
Strength of deep spinal muscles | 3 minutes
  Assessement will be with "Stabilizer".
Mobility | 5 minutes
  Prosthesis Evaluation Questionnaire (PEQ) was designed as a self-report visual analog scale style questionnaire with scores expressed in millimeters (0-100 mm). PEQ was previously translated to Turkish language, and it was proven to be valid and reliable. The questions of the PEQ are organized into nine functional domain scales, each reflecting a major area of concern for persons with amputations, such as "mobility". Each domain scale can be used and scored independent of the others. All subscales are scored between 0 and 100 (for example, in mobility subscale higher scores indicate higher mobility). In mobility subscale there are 13 questions. The minimum value that can be obtained as a result of the evaluation is 0 (minimum mobility), the maximum value is 130 (maximum mobility).

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Erbahceci, Prof, Study Chair — Hacettepe University; Senay Cerezci Duygu, MSc, Study Director — Baskent University
Locations (1):
- Baskent University, Ankara, Etimesgut, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No